CLINICAL TRIAL: NCT01403532
Title: Efficacy and Safety of Human Chorionic Gonadotropin (HCG) and Follicle Stimulating Hormone (FSH) in the Treatment of Hypogonadotropic Hypogonadism
Brief Title: Sequential Therapy for Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiao-Ying Li, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD005
Record Dates: First submitted 2011-02-01; First posted 2011-07-27 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Hypogonadotropic Hypogonadism; Kallmann Syndrome
Keywords: Hypogonadotropic Hypogonadism; Kallmann Syndrome; LH; FSH
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional (Active Comparator)
  Interventions: Drug: Traditional intervention for HH using HCG and FSH
- Sequential (Experimental)
  Interventions: Drug: Sequential intervention for HH using HCG and FSH
- Sequential Plus (Experimental)
  Interventions: Drug: Sequential intervention for HH using HCG and FSH plus zinc

INTERVENTIONS:
Drug: Traditional intervention for HH using HCG and FSH — Human chorionic gonadotropin(HCG),2000U,im,2 times/week, one year and a half; Follicle stimulating hormone(FSH),75U, im, 3 times/week, one year;
  Other Names: Tranditional
  Arms: Traditional
Drug: Sequential intervention for HH using HCG and FSH — Human chorionic gonadotropin,2000U,im, 2 times/week, one and half a year Follicle stimulating hormone,75U,im,3 times/week, every other three months
  Other Names: Sequential
  Arms: Sequential
Drug: Sequential intervention for HH using HCG and FSH plus zinc — Human chorionic gonadotropin,2000U,im,2 times/week, one year and a half Follicle stimulating hormone,75U, im, 3 times/week, every other three months Zinc gluconate 20mg,P.O, twice daily
  Other Names: Sequential plus
  Arms: Sequential Plus

SUMMARY:
The traditional therapy for induction of spermatogenesis in male hypogonadotropic hypogonadism requires both HCG and human menopausal gonadotropin (HMG) or FSH until pregnancy occurs. Because of the high cost of hMG or FSH preparations and poor compliance, the investigators raise a new sequential therapeutic approach which can make the treatment more economic and tolerable. The zinc supplement will be also evaluated in patients in this study. This randomized, parallel, open, and multi-center study will compare the efficacy of traditional therapy with new therapy and evaluate the safety of the new protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical hypogonadotropic hypogonadism
* Hormonal levels: Testosterone < 1.8ng/ml, LH < 2-3 mIU/mL and FSH < 2-3 mIU/mL
* Infantile testis
* Delayed bone age
* Normal testing of the anterior pituitary gland

Exclusion Criteria:

* Prior therapy with HMG or FSH
* Severe dysfunction of live and kidney
* Cryptorchidism or no response to HCG stimulation experiment (Testosterone < 1.8ng/ml after HCG stimulation)
* Another pituitary hormonal deficiency
* Hypergonadotropic hypogonadism
* With abnormal karyotype

Ages: 16 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sperm density ≥1,000,000/ml | One and a half year
  The sperm will be counted as equal or more than 1,000,000/ml under microscope for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ying Li, MD,PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Rui Jin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang M, Tong G, Liu Y, Mu Y, Weng J, Xue Y, Luo Z, Xue Y, Shi L, Wu X, Sun S, Zhu Y, Cao Y, Zhang J, Huang H, Niu B, Li H, Guo Q, Gao Y, Li Z, Ning G, Zhu D, Li X; HHIS Study Group. Sequential Versus Continual Purified Urinary FSH/hCG in Men With Idiopathic Hypogonadotropic Hypogonadism. J Clin Endocrinol Metab. 2015 Jun;100(6):2449-55. doi: 10.1210/jc.2014-3802. Epub 2015 Mar 31. PMID 25825944